CLINICAL TRIAL: NCT05564299
Title: Impact of a Rapid Test for Gonorrhea and Chlamydia on the Clinical Management of Urethritis and Cervicitis in a Sexual Health Clinic
Brief Title: Rapid Diagnostic Assay for Gonorrhea and Chlamydia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Sexually Transmitted Diseases Association (Unknown)
Responsible Party: Principal Investigator, Ingrid V. Bassett, MD, MPH, Associate Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022P002099
Record Dates: First submitted 2022-09-15; First posted 2022-10-03 (Actual); Results first posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Urethritis; Cervicitis; Sexually Transmitted Infections
MeSH Terms: conditions — Urethritis; Uterine Cervicitis; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard of Care (No Intervention): Point-of-care gram stain
- Rapid STI Test (Experimental)
  Interventions: Diagnostic Test: Rapid 30-minute Desktop Assay

INTERVENTIONS:
Diagnostic Test: Rapid 30-minute Desktop Assay — Participants will undergo routine evaluation and specimen collection per current clinic protocols. Specimens will be processed by the rapid 30-minute desktop assay. Concurrently, specimens will be used to create a point-of-care gram stain, to be read by the clinician following the clinical encounter.
  Treatment for urethritis and cervicitis will be provided based on results from the 30-minute assay.
  Specimens will also be plated for Gonorrhea culture and sent to the Massachusetts Department of Public Health for additional Gonorrhea and Chlamydia polymerase chain reaction testing, as per clinic protocols.
  Arms: Rapid STI Test

SUMMARY:
This study is a pilot randomized controlled trial evaluating the use of either a) rapid 30-minute desktop assay or b) point-of-care gram stain (current standard of care) to guide the clinical management of patients with symptomatic urethritis or cervicitis evaluated in the Massachusetts General Hospital Sexual Health Clinic. Patients presenting with symptoms of urethritis or cervicitis and meeting inclusion criteria will be randomized to have diagnostic specimens tested during the clinical encounter using either the 30-minute desktop assay or point-of-care gram stain. Patients randomized to the intervention arm of the study will also have a gram stain created, which will be held for interpretation by the clinician following the clinical encounter. Patients will not be followed longitudinally. Recruitment will conclude when 100 participants enroll in the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Presenting with symptoms of acute urethritis or cervicitis
* Willing to provide urine or additional vaginal swab specimen

Exclusion Criteria:

* Younger than 18 years old
* Presenting with symptoms not consistent with urethritis or cervicitis
* Unwilling or unable to provide urine or vaginal swab specimen
* Pregnant
* Contact of index patients with Gonorrhea or Chlamydia
* Known exposure to Gonorrhea or Chlamydia
* Reporting concurrent symptoms at a non-genital site
* Suspected or confirmed to have Monkeypox

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid V. Bassett, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Rapid STI Test: 30-minute point of care test for gonorrhea/chlamydia
Period: Overall Study
Arm/Group | Standard of Care | Rapid STI Test
Started | 49 | 49
Completed | 49 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Rapid STI Test | Total
Number analyzed (Participants) | 49 | 49 | 98
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 28 [24 to 35] | 31 [26 to 39] | 29.5 [25 to 39]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Cisgender male | 34 | 28 | 62
  Cisgender female | 13 | 19 | 32
  Transgender/nonbinary | 1 | 2 | 3
  Other | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 7 | 17
  Not Hispanic or Latino | 30 | 35 | 65
  Unknown or Not Reported | 9 | 7 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 5 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 12 | 20
  White | 26 | 18 | 44
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Mean Antibiotic Days of Therapy (DOT) Administered Per Patient With Symptomatic Urethritis or Cervicitis
Description: The investigators will compare the mean antibiotic days of therapy (DOT) administered per patient at the time of initial ciinical visit when evaluated with either point-of-care gram stain or rapid 30-minute desktop test.
Time Frame: Day 1
Measure: Median (Inter-Quartile Range); unit: Antibiotic days of therapy (DOT)
Arm/Group | Standard of Care | Rapid STI Test
Number analyzed (Participants) | 49 | 49
Antibiotic days of therapy (DOT) | 7 [0 to 8] | 1 [0 to 7]
Statistical Analysis 1: Comparison: Standard of Care vs Rapid STI Test; Wilcoxon rank sum test; Test type: Other; p = 0.053, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Participant Visit Duration
Description: The investigators will compare visit duration between participants randomized to the point-of-care test and those to the 30-minute desktop test. Participant visit duration will be calculated as the difference between when the participant enters the exam room and when they check out of the clinic, in minutes.
Time Frame: Day 1
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Standard of Care | Rapid STI Test
Number analyzed (Participants) | 49 | 49
Minutes | 57 [45 to 69] | 87 [72 to 97]

3. Secondary Outcome: Sample Processing Time
Description: The investigators will compare the time taken to process clinical specimen using either the point-of-care gram stain or rapid 30-minute desktop test. The provider processing the samples will record the start and end times on a time sheet, and the sample processing time will be calculated as the difference between those entries, in minutes.
Time Frame: Day 1
Population: This outcome measure was not collected. At the start of the study, it was determined that staff would not be able to accurately document the sample processing time in the clinical context, as stopping between sample processing and running or reading the test was not feasible and disrupted the providers' workflow, thus potentially altering the outcomes of other process measures. This change was made after the start of the study but not amended specifically in the protocol.
Arm/Group | Standard of Care | Rapid STI Test
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Time to Result
Description: The investigators will compare time from specimen collection to availability of test result between the point-of-care gram stain or rapid 30-minute desktop test. Providers will record time of specimen collection and time of result (for point of care gram stain), time of result for the rapid desktop platform will be extracted from the platform; time to result will be calculated as the difference between those times, in minutes.
Time Frame: Day 1
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Standard of Care | Rapid STI Test
Number analyzed (Participants) | 49 | 49
Minutes | 6.5 [5 to 9] | 34 [33 to 36]

5. Secondary Outcome: Test-concordant Antibiotic Use for Gonorrhea
Description: Proportion of participants in each arm who recevied gonorrhea-active antibiotics if PCR-based testing (rapid test or MDPH) was positive for gonorrhea, or who did not receive gonorrhea-active antibiotics if PCR-based testing (rapid test or MDPH) was negative for gonorrhea
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Rapid STI Test
Number analyzed (Participants) | 49 | 49
Participants | 41 | 46

6. Secondary Outcome: Diagnosis-concordant Antibiotic Use for Gonorrhea
Description: Proportion of participants in each arm who were prescribed an antibiotic with activity against gonorrhea on the day of clinic visit, either for a positive test result or for a clinical syndrome for which the antibiotics are indicated (e.g., a clinical diagnosis of pelvic inflammatory disease, a diagnosis of non-gonococcal urethritis) as determined by study PI; or who were not prescribed an antibiotic with activity against gonorrhea on the day of clinic visit in the absence of a positive test result for gonorrhea or clinical syndrome for which the antibiotics are indicated.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Rapid STI Test
Number analyzed (Participants) | 49 | 49
Participants | 43 | 48

7. Secondary Outcome: Proportion of Participants With Invalid or Unavailable Point of Care Gram Stain or Rapid STI Test Results
Description: The proportion of point of care gram stain results (control arm) or rapid test results (intervention arm) that were unavailable or invalid (unable to be read or provided an error message) at the time of the clinic visit.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Rapid STI Test
Number analyzed (Participants) | 49 | 49
Participants | 4 | 0

8. Other Pre Specified Outcome: Clinic Provider Perspectives on Rapid STI Testing
Description: Clinic provider perspectives will be elicited during a focus group discussion at the conclusion of the clinical study.
Time Frame: at study completion: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Standard of Care | Rapid STI Test
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 0/49 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-30): https://cdn.clinicaltrials.gov/large-docs/99/NCT05564299/Prot_SAP_000.pdf